CLINICAL TRIAL: NCT04022733
Title: A Double-blind, Randomized Study to Compare the Remifentanil Requirements in Deep Versus Moderate Neuromuscular Blocks During the Surgical Pleth Index-guided Analgesia in Patients Undergoing General Anesthesia for Laparoscopic Herniorrhaphy
Brief Title: Remifentanil in Deep vs Moderate Neuromuscular Blocks During Surgical Pleth Index-guided Anesthesia for Laparoscopic Herniorrhaphy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ajou University School of Medicine (Other)
Responsible Party: Principal Investigator, Ji Eun Kim, Assistant professor, Ajou University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: AJIRB-MED-THE-19-056
Record Dates: First submitted 2019-07-15; First posted 2019-07-17 (Actual); Results first posted 2022-03-15 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Hernia Abdominal Wall
MeSH Terms: conditions — Hernia, Abdominal

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Moderate NMB group (Placebo Comparator)
  Interventions: Drug: Moderate neuromuscular block
- Deep NMB group (Experimental)
  Interventions: Drug: Deep neuromuscular block

INTERVENTIONS:
Drug: Moderate neuromuscular block — maintaining of moderate neuromuscular block (train-of-four count 1-2) during surgery, reversal using neostigmine 50 ug/kg and glycopyrrolate 10 ug/kg
  Arms: Moderate NMB group
Drug: Deep neuromuscular block — maintaining of deep neuromuscular block (posttetanic count 1-2) during surgery, reversal using sugammadex 4 mg/kg based on actual body weight
  Arms: Deep NMB group

SUMMARY:
The primary purpose of this study is to compare the remifentanil requirements in deep versus moderate neuromuscular blocks during the surgical pleth index -guided anesthesia in patients undergoing laparoscopic herniorrhaphy.

ELIGIBILITY:
Inclusion Criteria:

* laparoscopic hernia repair

Exclusion Criteria:

* patients refusal, hyperbilirubinemia, chronic pain, opioid abuse, infection, and peripheral disease

Ages: 19 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2019-10-30 (Actual); Primary Completion 2021-08-03 (Actual); Study Completion 2021-08-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Ajou University School of Medicine, Suwon, Gyeonggido, South Korea

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Moderate NMB Group | Deep NMB Group
Started | 67 | 67
Completed | 64 | 64
Not Completed | 3 | 3
Not completed — conversion to open surgery | 3 | 2
Not completed — bradycardia | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Moderate NMB Group | Deep NMB Group | Total
Number analyzed (Participants) | 64 | 64 | 128
Age, Continuous [Median (Inter-Quartile Range); unit: year] | 63 [54 to 70] | 65 [51 to 75] | 63.5 [52.8 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 11
  Male | 58 | 59 | 117
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 64 | 64 | 128
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  South Korea | 64 | 64 | 128

OUTCOME MEASURES:

1. Primary Outcome: Remifentanil Infusion Rate
Description: remifentanil infusion using target effect-site concentration to achieve an surgical pleth index of range between 25 and 50
Time Frame: from pneumoperitoneum to removal of laparoscope, an average of 30 minutes
Measure: Mean (Inter-Quartile Range); unit: µg/kg/min
Arm/Group | Moderate NMB Group | Deep NMB Group
Number analyzed (Participants) | 64 | 64
µg/kg/min | 0.103 [0.075 to 0.143] | 0.073 [0.056 to 0.097]

ADVERSE EVENTS:
Time Frame: from the start of anesthesia induction until discharge of post-anesthesia care unit, an average of 130 minutes
Description: Complications regarding deep NMB or sugammadex use
Arm/Group | Moderate NMB Group | Deep NMB Group
All-Cause Mortality (participants affected / at risk) | 0/67 | 0/67
Serious Adverse Events (participants affected / at risk) | 0/67 | 0/67
Other Adverse Events (participants affected / at risk) | 0/67 | 0/67

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-01-18): https://cdn.clinicaltrials.gov/large-docs/33/NCT04022733/Prot_000.pdf
  • Statistical Analysis Plan (2022-01-18): https://cdn.clinicaltrials.gov/large-docs/33/NCT04022733/SAP_001.pdf